CLINICAL TRIAL: NCT01497067
Title: Long Term Safety Follow-up for Subjects Previously Implanted With the ACRYSOF® CACHET® Phakic Lens in Clinical Studies C-02-23, C-02-40, C-03-21 and C-05-57
Brief Title: Long Term Safety Protocol for the AcrySof CACHET Phakic Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-09-043
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Myopia
Keywords: Phakic Lens; Intraocular Lens (IOL)
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CACHET (Experimental): ACRYSOF CACHET Phakic Lens (L-series) previously implanted
  Interventions: Device: ACRYSOF CACHET Phakic Lens (L-series)

INTERVENTIONS:
Device: ACRYSOF CACHET Phakic Lens (L-series) — Intraocular lens for the treatment of moderate to high myopia
  Other Names: AcrySof Angle-Supported Phakic Lens

SUMMARY:
The purpose of this long term safety study is to estimate the annualized endothelial cell loss (ECL) rate (for up to 10 years following date of implantation) of subjects previously implanted with the ACRYSOF CACHET Phakic Intraocular Lens (L-series) from precursor clinical studies C-02-23, C-02-40, C-03-21 and C-05-57.

DETAILED DESCRIPTION:
Subjects previously enrolled in protocols C-02-23 (NCT00726024), C-02-40 (NCT00727805), C-03-21 (NCT00726297), and C-05-57 (NCT00727688) who received an L-series lens either in the first eye or second eye (including those who were explanted) were enrolled in this open-label, non-randomized, non-controlled, extension study in which they attended postoperative visits for up to 10 years following the date of implantation. Subjects could enroll in the study at any time, thus the Entrance Visit may have coincided with any visit (Year 4 to Year 10).

ELIGIBILITY:
Inclusion Criteria:

* Previously implanted with an ACRYSOF CACHET Phakic Lens (L-Series) from clinical studies C-02-23, C-02-40, C-03-21 and C-05-57 and eligible for continued follow-up (i.e., exited from the previous study).
* Able to understand and sign a statement of informed consent.
* Willing and able to complete the yearly postoperative study visits.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Project Lead, Surgical, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects at 20 investigative sites located in the US, 9 investigative sites located in the European Union, and 5 investigative sites located in Canada.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Period: Overall Study
Arm/Group | CACHET
Started | 657
Completed | 575
Not Completed | 82
Not completed — Lost to Follow-up | 56
Not completed — Adverse Event | 3
Not completed — Patient decision unrel to Adverse Event | 10
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Arm/Group | CACHET
Number analyzed (Participants) | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 448
  Male | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 597
  Black or African American | 14
  Asian | 34
  Hispanic | 3
  Multi-racial | 1
  Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Central Endothelial Cell Density (All Eyes)
Description: A microscope was used to photograph corneal endothelial cells (cells on the back of the cornea). Three images at the center of the cornea were obtained and sent to a central reading center for analysis. All recorded data from images were used in the analysis. A higher value for density represents a healthier cornea.
Time Frame: Year 4 to Year 10 postoperative from previous study (C-02-23, C-02-40, C-03-21, and C-05-57)
Population: All subjects enrolled in the study (Safety Analysis). Some subjects were implanted in both eyes and therefore 2 eyes were enrolled.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | CACHET
Number analyzed (Participants) | 657
Number analyzed (eyes) | 1123
cells/mm^2
  Year 4: number analyzed (Participants) | 69
  Year 4: number analyzed (eyes) | 80
  Year 4 | 2654.0 (354.6)
  Year 5: number analyzed (Participants) | 259
  Year 5: number analyzed (eyes) | 446
  Year 5 | 2639.0 (324.2)
  Year 5.5: number analyzed (Participants) | 65
  Year 5.5: number analyzed (eyes) | 81
  Year 5.5 | 2633.0 (357.6)
  Year 6: number analyzed (Participants) | 371
  Year 6: number analyzed (eyes) | 629
  Year 6 | 2551.0 (362.3)
  Year 6.5: number analyzed (Participants) | 310
  Year 6.5: number analyzed (eyes) | 532
  Year 6.5 | 2524.7 (360.6)
  Year 7: number analyzed (Participants) | 490
  Year 7: number analyzed (eyes) | 803
  Year 7 | 2504.9 (365.8)
  Year 7.5: number analyzed (Participants) | 449
  Year 7.5: number analyzed (eyes) | 726
  Year 7.5 | 2497.1 (364.7)
  Year 8: number analyzed (Participants) | 567
  Year 8: number analyzed (eyes) | 884
  Year 8 | 2465.0 (384.2)
  Year 8.5: number analyzed (Participants) | 492
  Year 8.5: number analyzed (eyes) | 780
  Year 8.5 | 2457.7 (363.0)
  Year 9: number analyzed (Participants) | 561
  Year 9: number analyzed (eyes) | 856
  Year 9 | 2409.6 (388.4)
  Year 9.5: number analyzed (Participants) | 544
  Year 9.5: number analyzed (eyes) | 825
  Year 9.5 | 2399.3 (387.9)
  Year 10: number analyzed (Participants) | 575
  Year 10: number analyzed (eyes) | 872
  Year 10 | 2377.5 (398.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment until study exit for an individual duration up to 6 years based on time of enrollment.
Description: Adverse Events (AE) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. This analysis population includes all subjects enrolled in the study. Number at risk for ocular adverse events is presented with unit eyes.
Groups:
- CACHET - Ocular: All eyes previously implanted with ACRYSOF CACHET Phakic Lens (L-series)
- CACHET - Systemic: All subjects previously implanted with ACRYSOF CACHET Phakic Lens (L-series)
Arm/Group | CACHET - Ocular | CACHET - Systemic
All-Cause Mortality (participants affected / at risk) | 0/1123 | 3/657
Serious Adverse Events (participants affected / at risk) | 276/1123 | 24/657
Other Adverse Events (participants affected / at risk) | 0/1123 | 0/657
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CACHET - Ocular (N=1123) | CACHET - Systemic (N=657)
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 3 | 0
Cataract (Eye disorders) | 20 | 0
Cataract cortical (Eye disorders) | 8 | 0
Cataract nuclear (Eye disorders) | 66 | 0
Cataract subcapsular (Eye disorders) | 10 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0
Corneal endothelial cell loss (Eye disorders) | 99 | 0
Corneal oedema (Eye disorders) | 1 | 0
Exophthalmos (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 6 | 0
Iris adhesions (Eye disorders) | 88 | 0
Iris atrophy (Eye disorders) | 2 | 0
Iris disorder (Eye disorders) | 2 | 0
Lens discolouration (Eye disorders) | 2 | 0
Lens dislocation (Eye disorders) | 1 | 0
Lenticular opacities (Eye disorders) | 5 | 0
Macular oedema (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 4 | 0
Open angle glaucoma (Eye disorders) | 5 | 0
Pupillary deformity (Eye disorders) | 6 | 0
Retinal degeneration (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 3 | 0
Retinal tear (Eye disorders) | 2 | 0
Visual acuity reduced (Eye disorders) | 11 | 0
Accidental death (General disorders) | 0 | 1
Device dislocation (General disorders) | 7 | 0
Eye complication associated with device (General disorders) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 2
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Intraocular pressure increased (Investigations) | 11 | 0
Visual acuity tests abnormal (Investigations) | 3 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Visual field defect (Nervous system disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cataract operation (Surgical and medical procedures) | 2 | 0
Corneal operation (Surgical and medical procedures) | 5 | 0
Eye operation (Surgical and medical procedures) | 1 | 0
Glaucoma surgery (Surgical and medical procedures) | 2 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1
Intra-ocular injection (Surgical and medical procedures) | 1 | 0
Intraocular lens extraction (Surgical and medical procedures) | 119 | 0
Intraocular lens implant (Surgical and medical procedures) | 64 | 0
Intraocular lens repositioning (Surgical and medical procedures) | 2 | 0
Iridotomy (Surgical and medical procedures) | 3 | 0
Iris operation (Surgical and medical procedures) | 2 | 0
Keratomileusis (Surgical and medical procedures) | 10 | 0
Knee operation (Surgical and medical procedures) | 0 | 1
Lens extraction (Surgical and medical procedures) | 1 | 0
Retinal laser coagulation (Surgical and medical procedures) | 7 | 0
Retinal operation (Surgical and medical procedures) | 1 | 0
Retinopexy (Surgical and medical procedures) | 4 | 0
Scleral buckling surgery (Surgical and medical procedures) | 1 | 0
Trabeculectomy (Surgical and medical procedures) | 2 | 0
Trabeculoplasty (Surgical and medical procedures) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 3 | 0
Hypertension (Vascular disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT01497067/SAP_000.pdf
  • Study Protocol (2013-04-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT01497067/Prot_001.pdf